CLINICAL TRIAL: NCT02771600
Title: Feasibility, Acceptability and Satisfaction of a New Device (Buzzy®) for Pediatric Procedural Pain and Anxiety Management During Needle-Related Procedures: A Pilot Study.
Brief Title: Pilot Study of a New Device (Buzzy®) for Procedural Pain Relief During Needle-Related Procedures in Paediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Toronto-Dominion Bank of Canada Funds for Clinical Research projects. (Unknown)
Responsible Party: Principal Investigator, Ariane Ballard, Doctoral student, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4137
Record Dates: First submitted 2016-05-09; First posted 2016-05-13 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Autoimmune Rheumatologic Disease; Immune Deficiency; Pain Due to Certain Specified Procedures; Child/Adolescent Problems
Keywords: Procedural pain; Procedural anxiety; Pediatrics; Needle-related procedures
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Pain, Procedural | interventions — Maxilene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buzzy (Experimental): Just before the needle-related procedure, the Buzzy®, combining an ice pack and vibration integrated to a plastic bee, will be applied 5 cm above the needle insertion site and will be maintained in place throughout the painful procedure.
  Interventions: Device: Buzzy
- Standard Care (Maxilene) (Active Comparator): Maxilene topical anaesthetic cream will be applied 30 minutes before the needle-related procedure on the insertion site
  Interventions: Drug: Topical anaesthetic cream

INTERVENTIONS:
Device: Buzzy — See arm description
  Arms: Buzzy
Drug: Topical anaesthetic cream — See arm description
  Other Names: Maxilene
  Arms: Standard Care (Maxilene)

SUMMARY:
Needle-related procedures are the most important source of pain and anxiety in pediatric patients. Consequently, needle-phobia and anxiety are common in children with auto-immune disease and immune deficiency and may be barriers to adherence in treatment. The use of a non-pharmacological and easy-to-use approach, like the Buzzy® device, could be an alternative or adjuvant for the management of procedural pain and anxiety of these children during needle-related procedures.

This study aims to determine the feasibility, acceptability and satisfaction of the Buzzy® device for procedural pain and anxiety relief of immunology-rheumatology patients undergoing needle-related procedures. The investigators will compare the Buzzy® device with an anaesthetic cream (Maxilene®) during needle-related procedures. The investigators also plan to assess feasibility outcomes and satisfaction of the nurses and the children with the use of the Buzzy® device. This pilot study should refine or modify the research methodology and improve the intervention being piloted before it's efficacy will be verified within a larger scale-study.

The investigators strongly believe that the use of the Buzzy® device in immunology rheumatology department could optimise procedural pain and anxiety management. Since most of the treatments administered for auto-immune diseases and immune deficiency diseases are through subcutaneous or intramuscular injections, pain and anxiety management using non-pharmacological and/or pharmacological interventions should be prioritized. Given this knowledge, the investigators feel that this pilot study has the potential to contribute to pain and anxiety management of children undergoing needle-related procedures.

DETAILED DESCRIPTION:
Rationale: Procedural pain and anxiety relief of needle-related procedures is a major concern for nurses working with Immunology-Rheumatology patients. Treatments for most autoimmune diseases and immune deficiencies diseases are administrated by subcutaneous or intramuscular injections and these children will go through countless needle-related procedures for a long period of their life. Procedural pain and anxiety generates consequences which may be physiological, psychological and emotional. Since it is impossible to completely control pain and anxiety experienced by pediatric patients during painful procedures, non-pharmacological and/or pharmacological interventions should be part of the interventions to provide comfort to children. Interventions to decrease physical and emotional impacts of needle-related procedures should be an integral part of nursing activities. Most of pain and anxiety management methods available for children require much time of staff, which represents barriers to their implantation among nursing interventions. Use of a rapid and easy-to-use non-pharmacological intervention could overcome these constraints and optimise pain and anxiety relief in children. Investigators believe that the Buzzy® device, combining cold and vibration, could be an efficient way to improve pain and anxiety management during needle-related procedures. To date, no studies have focused on the efficacy of this device on pediatric immunology-rheumatology patients.

Objective: To assess the feasibility, acceptability and satisfaction of a new device (Buzzy®) combining the effect of cold and vibration, for procedural pain relief and anxiety during needle-related procedures in pediatric immunology-rheumatology patients.

Methods. Design: This study is a pilot study of a two-group randomized controlled trial (RCT). Setting: Immunology-Rheumatology clinic of the CHU Sainte-Justine's (Montreal). Inclusion criteria: We will include children: a) between the ages of 4 and 17 years old; b) visiting the Immunology-Rheumatology Clinic for a follow-up; c) who require a s/c injection or IM injection or venipuncture or IV catheter insertion; d) who understand French or English; e) who have at least one parent who understand, read and talk French or English. Exclusion criteria: We will exclude children: a) who have a diagnosed neuro-cognitive disability that precludes patients from assenting and participating to the study, b) who have the inability to self-report pain. Sample size: We expect to recruit 100 participants for this pilot study (50 participants per group). Allocations: According to a randomized list, patients will be allocated to one of the study group: a) Experimental group: Just before the needle-related procedure, the Buzzy® device, combining an ice pack and vibration integrated to a plastic bee, will be applied 5 cm above the needle insertion site and will be maintained in place throughout the painful procedure; or b) Control group: Maxilene® topical anaesthetic cream will be applied 30 minutes before the needle-related procedure on the insertion site. Primary outcomes: Post-procedural pain and it will be measured with the Faces Pain Scale-Revised (FPS-R) (4-12 years old) and the Numerical Pain Rating Scale (NPRS) (>12 years old). Secondary outcomes: Post-procedural anxiety and it will be measured with the Procedure Behavior Check List (PBCL). We will also assess the satisfaction of nurses and children regarding the Buzzy® device. Satisfaction will be measured using questionnaires previously developed by investigators. The principal feasibility outcomes will be the recruitment rates, the refusal rate, the needle-related procedure rate and the time of the procedure. Study times periods: Four study times periods are planned: T-0: before randomization; T-1: 5 min. before the needle-related procedure (pre-procedural pain and pre-procedural anxiety); T-2: immediately after the needle-related procedure (post-procedural pain and post-procedural anxiety); T-3: 15 min. after the needle-related procedure (satisfaction and feasibility outcomes). Data analysis: Descriptive statistics will be used for group characteristics. Quantitative multivariate analysis will be performed to compare both groups for pre- and post-procedural pain and anxiety. Descriptive statistics will be used for report on satisfaction and feasibility outcomes. ANCOVA will be used on covariate to increase statistical power.

Relevance: This pilot study will assess the effects of a new device on pain and anxiety level of immunology-rheumatology patients during needle-related procedure and will test feasibility of the study design as well as acceptability on the new distraction device by patients and nurses. This study will refine the research methodology and improve the intervention being piloted for a future large-scale study.

ELIGIBILITY:
Inclusion Criteria: We wil include children:

* Between the ages of 4 and 17 years old
* Who have a follow-up at the Immunology-Rheumatology Clinic
* Who require a s/c injection or IM injection or venipuncture or IV catheter insertion
* Who understand and speak French or English
* Who have at least one parent who understand, read and talk French or English

Exclusion Criteria: We will exclude children:

* With a diagnosed neuro-cognitive disability that precludes patients from assenting and participating to the study
* Who are unable to self-report pain

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Post-procedural Pain | T-2: Immediately after the needle-related procedure
  To assess the pain intensity after the needle-related procedure. Measure : Faces Pain Scale-Revised (4-12 years old), Numerical Rating Pain Scale (NRPS) (>12 years old).

SECONDARY OUTCOMES:
Anxiety level | T-1: 5 min. before the needle-related procedure, T-2: Immediately after the needle-related procedure
  To assess the anxiety level during all the time periods of the study. Measures: Procedure Behaviour Check List (PBCL)
Satisfaction of the parents, children and nurses | T-3: 15 min. after the needle-related procedure
  To assess satisfaction of nurses and children regarding the Buzzy® device. Measures : Questionnaires previously developed by investigators.
Process time of the needle-related procedure | T-2: Immediately after the needle-related procedure
  To assess the feasibility of this study. Measures: Clinical data.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Le May, PhD, Principal Investigator — CHU Ste-Justine's
Locations (1):
- CHU Ste-Justine's, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No